CLINICAL TRIAL: NCT06601556
Title: Evaluation of Psychiatric Problems Among Thalassemic Children in Assuit University Children Hospital
Brief Title: Psychiatric Problems in Thalassemic Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Amary, Resident doctor, Assiut University
Other Study IDs: Psychiatric in thalassemia
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psychiatric and Thalassemia; Psychiatry and Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Aims of the study :

1. Assessment the prevalence of psychiatric problems in thalassemic children .
2. Assessment the prevalence of cognitive problems in thalassemic children .
3. Determine factors associated with psychiatric and cognitive problems in thalassemic children .

Sociodemographic information, other associated factors , CBCL (Child Behaviour Check List) and Children's Sleep Habits Questionnaire will be collected by thalassemic child's caregiver interview at Assiut university ,Children hospital , pediatric hematology unit .

Raven´s Colored Progressive Matrices will be solved by thalassemic patient at Assiut university , Children hospital , pediatric hematology unit .

DETAILED DESCRIPTION:
Beta-thalassemia is a chronic and genetically determined hematological disorder characterized by severe hemolytic anemia as a result of deficient synthesis of β chains of hemoglobin.

β-Thalassemia major is considered the commonest hemoglobinopathy in the Mediterranean area particularly Egypt with an estimated carrier rate of 9-10.2 % . From about registered β-thalassemia cases ; 95% of them are β-thalassemia major, and 5% are thalassemia intermediate.

It demands frequent blood transfusions to maintain life, while haemosiderosis and other complications of the disease require a continuous and distressing treatment regimen that includes parenteral iron chelation treatment and regular medical supervision.

The drawbacks of the disease in many aspects of life become strongly evident during the school age when children ask for independence . It has been related with psychosocial aspect and a significant negative effect on areas of school functioning because of the likelihood of physical deformity, growth retardation and delayed puberty besides the difficulty of management (such as regular transfusion and time-consuming iron chelation treatment) Social stigma associated with having thalassaemia have significant psychosocial and emotional impact on patients and their families(3) , so The affected children become more liable to emotional, social, psychological and behavioural problems .

No available studies about psychiatric problems among thalassemic children in Egypt . Also study that were conducted in the age < 12 years are few .

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 6 to < 12 years.

Exclusion Criteria:

1. Patients who had bone marrow transplant and were cured of thalassemia .
2. Neurological illness preventing them from expressing themselves and not able to communicate well

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Thalassemic patients between 6 and 12 years old
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
• Assessment the prevalence of psychiatric problems in thalassemic children | One year
  By using CBCL (Child Behaviour Check List) is a questionnaire based standardized tool used for assessing behavioural problems(6) . CBCL for school aged children (6-18 years) in local language is filled by the primary caregivers/parents after obtaining written consent . It contains 113 questions categorized into eight domains which are anxious/depressed, withdrawn, somatic complaints, social problems, thought problems, attention problems, rule breaking behaviour and aggressive behaviour.(7)

SECONDARY OUTCOMES:
• Determine factors associated with psychiatric and cognitive problems in thalassemic children . • Assessment the prevalence of cognitive problems in thalassemic children | One year
  By using Raven´s Colored Progressive Matrices (CPM)-Sets A, AB, B standardized for the population between 6 and 11 years old, comprises 36 items, in which the subject is required to indicate the correct target among six alternatives. Grouped into three sets (A, AB, B) of 12 items in each one, the CPM solving requires different abilities, namely: A Series, requiring visuo-perceptual ability; AB Series, symmetric ability; and B Series, conceptual and analogic thought abilities
  Associated factor by sociodemographic data Name, age, gender, residence (urban or rural and live with family or extended family) and education (student or not , and if not the last degree) and socioeconomic level by by Fahmy and El Sherbini Socio- economic status (SES) scale.the scale consist of 7 domains with total score 84, each domain contain many items that collectively it can measure the socioeconomic status of the family

CONTACTS AND LOCATIONS:
Overall Officials: Gellan Gellan Karamallah, Lecturer, Study Director — Assiut University; Khaled Khaled Elsayh, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided